CLINICAL TRIAL: NCT05126134
Title: Psychological Vulnerabilities and Transgender Adolescents: A Descriptive Epidemiology Study
Acronym: VATED
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0385
Record Dates: First submitted 2021-11-03; First posted 2021-11-18 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Gender Dysphoria, Adolescent
Keywords: mental disorders
MeSH Terms: conditions — Gender Dysphoria; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adolescents followed for gender dysphoria: The data collection by the examiner takes place during a single interview centered around the child's completion of a semi-structured questionnaire: the Kiddie Schedule for Affective Disorders and Schizophrenia. The child is interviewed alone and then with an accompanying parent.
  Interventions: Diagnostic Test: KSADS (Kiddie Schedule for Affective Disorders and Schizophrenia)

INTERVENTIONS:
Diagnostic Test: KSADS (Kiddie Schedule for Affective Disorders and Schizophrenia) — completion of the semi-structured questionnaire: the KSADS (Kiddie Schedule for Affective Disorders and Schizophrenia). The duration is 1h30 to 2h

SUMMARY:
The number of adolescents engaging in a transidentity journey has been increasing rapidly over the last decade. However, the knowledge of the medical world concerning the specificities of these adolescents is still too little in France. The objective of this study is to refine the knowledge of the different health care providers who are brought to meet these adolescents. This research proposes to study more specifically the register of psychological vulnerabilities: to cite only a few examplesThese include disorders such as depression, anxiety disorders and eating disorders, all of which cause suffering and difficulties in everyday life. A better understanding of the presence or absence and the distribution of these different types of vulnerabilities among transgender adolescents would allow, among other things, to promote their their screening by health care providers. This better screening would allow doctors to physicians to offer targeted treatment for these disorders in parallel with the transition process. transition process.

ELIGIBILITY:
Inclusion Criteria:

* Be between 12 and 18 years old
* Be followed up at the gender consultation of the Toulouse University Hospital

Exclusion Criteria:

* Have not yet completed the first consultation on gender issues at the time of selection.
* Have only one last appointment with the gender consultation at the time of selection

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: adolescents receiving follow-up in a specialized consultation on gender dysphoria
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
list of diagnoses of mental disorders | enrollment
  description of the prevalence of psychiatric comorbidities present in adolescents receiving follow-up in a specialized consultation on gender dysphoria using Diagnostic and Statistical Manual of Mental Disorders 5

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Çabal-Berthoumieu, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Chu Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No